CLINICAL TRIAL: NCT05754645
Title: The PROMOTE Study, a Pilot: The Characterization of the Microbiome in Pregnancy and Prediction of Pregnancy Outcomes
Brief Title: The Microbiome in (Non-) Obese Pregnancy and Pregnancy Outcomes
Acronym: PROMOTE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Sam Schoenmakers, Principal Investigator, gynecologist-perinatologist, Erasmus Medical Center
Other Study IDs: NL80155.078.22/OZBS72.21318
Record Dates: First submitted 2023-01-24; First posted 2023-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity, Maternal; Pregnancy Complications; Gut Microbiota
MeSH Terms: conditions — Pregnancy in Obesity; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Vaginal sample (swab) Rectal sample (swab)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 110 women: 60 women with a BMI between 18,5-25 kg/m2, of which 10 preconceptional 60 women with a BMI > 30 kg/m2, of which 10 preconceptional
  Interventions: Other: Blood withdrawal

INTERVENTIONS:
Other: Blood withdrawal — venous punction with blood withdrawal Vaginal and rectal swab, done by patient itself
  Other Names: Vaginal/rectal swabs

SUMMARY:
This research aims to elucidate an underlying mechanism of maternal obesity induced pregnancy and longterm health complications for mothers and their offspring.

DETAILED DESCRIPTION:
With the increasing global prevalence of obesity, pregnancy problems related to maternal obesity are increasingly occurring. Microbial gut symbiosis plays an important role in health, with dysbiosis being associated with diseases such as obesity. Of interest are pregnancy, dietary patterns and pre- or probiotics that affect the composition of the gut microbiome. The microbiome itself can influence many physiological processes, such as immune responses (production of microbial products) and the nutrient-dependent one-carbon metabolism. It is hypothesized that gut dysbiosis, due to maternal obesity, during pregnancy can be considered an endogenous chronic stressor causing impaired immune response and carbon metabolism. Both processes result in excessive oxidative stress, detrimental to cell replication, differentiation and epigenetic programming of maternal and infant tissues. Together, these biological disturbances contribute to placental and vascular dysfunction, leading to an increased risk of preeclampsia or gestational diabetes mellitus. Vertical (during pregnancy) and horizontal (during delivery) transmission of gut dysbiosis from mother to newborn and epigenetic placental and foetal changes may ultimately lead to macrosomia and obesity in children. Therefore, the differences between the gut and vaginal microbiome, maternal and fetal immune responses and one-carbon metabolism in obese versus normal-weight pregnant women will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Predict study
* Preconceptional women who wish to become pregnant or pregnancy <13 weeks of gestational age.
* BMI > 30 kg/m2 or 18-25 kg/m2
* Understanding of Dutch in speaking and reading
* Willingness to give written informed consent

Exclusion Criteria:

* Age < 18 years and > 45 years.
* ≥13 weeks of gestational age
* Multiple pregnancy
* Smoking
* Gastro-intestinal diseases, heart diseases, liver, pancreas and kidney diseases.
* Use of antibiotics < 2 weeks before sampling
* Pre-existent diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This pilot study is embedded in the Rotterdam Periconceptional Cohort study (Predict study). The Predict study population includes preconceptional or pregnant women > 18 years and < 45 years old visiting the Erasmus MC and that are willing to participate. We will select the participants, that meet our undermentioned inclusion criteria, for our study from this cohort: 50 women with a BMI > 30 kg/m2 (cases) and 50 women with a BMI ranging 18-25 kg/m2 (controls) and their neonates.
  We will longitudinally sample first/2nd/3rd/postpartum, 100 women, in addition we will include 10 preconceptional women with BMI > 30 kg/m2 and 10 preconceptional women with BMI 18-25 kg/m2, these participants do not necessarily have to conceive a pregnancy in order to remain in the study (these women are part of the preconceptional Predict population).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Gut and vaginal microbiota | Preconceptional (up to 1 year before pregnancy)
  Composition of gut and vaginal microbiota derived by swab sampling, bacteriome profiles will be assessed by 16S ribosomal ribonucleic acid (16SrRNA) gene amplification sequencing (V6-V8). Sequences will be assigned to operational taxonomic units (OTUs).
Gut and vaginal microbiota | First trimester (between 7-12 weeks gestational age)
  Composition of gut and vaginal microbiota derived by swab sampling, bacteriome profiles will be assessed by 16SrRNA gene amplification sequencing (V6-V8). Sequences will be assigned to OTUs.
Gut and vaginal microbiota | Second trimester (between 22-25 weeks gestational age)
  Composition of gut and vaginal microbiota derived by swab sampling, bacteriome profiles will be assessed by 16SrRNA gene amplification sequencing (V6-V8). Sequences will be assigned to OTUs.
Gut and vaginal microbiota | Third trimester (between 30-32 weeks gestational age)
  Composition of gut and vaginal microbiota derived by swab sampling, bacteriome profiles will be assessed by 16SrRNA gene amplification sequencing (V6-V8). Sequences will be assigned to OTUs.
Gut and vaginal microbiota | Antepartum (during delivery)
  Composition of gut and vaginal microbiota derived by swab sampling, bacteriome profiles will be assessed by 16SrRNA gene amplification sequencing (V6-V8). Sequences will be assigned to OTUs.
Gut and vaginal microbiota | Postpartum (6-8 weeks post delivery)
  Composition of gut and vaginal microbiota derived by swab sampling, bacteriome profiles will be assessed by 16SrRNA gene amplification sequencing (V6-V8). Sequences will be assigned to OTUs.

SECONDARY OUTCOMES:
Gut virome | Preconceptional (up to 1 year before pregnancy)
  Composition of gut virome, obtained by a rectal swab
Gut virome | First trimester (between 7-12 weeks gestational age)
  Composition of gut virome, obtained by a rectal swab
Gut virome | Second trimester (between 22-24 weeks gestational age)
  Composition of gut virome, obtained by a rectal swab
Gut virome | Third trimester (between 30-32 weeks gestational age)
  Composition of gut virome, obtained by a rectal swab
Gut virome | Antepartum (during delivery)
  Composition of gut virome, obtained by a rectal swab
Gut virome | Postpartum (6-8 weeks post delivery)
  Composition of gut virome, obtained by a rectal swab
Maternal immune response | Preconceptional (up to 1 year before pregnancy)
  Responses of maternal immune system advanced oxidation protein products (AOPP)) measured in chloramine units per gram of protein (micromol/g) obtained by blood withdrawal and measured in the lab.
Maternal immune response | First trimester (between 7-12 weeks gestational age)
  Responses of maternal immune system advanced oxidation protein products (AOPP)) measured in chloramine units per gram of protein (micromol/g) obtained by blood withdrawal and measured in the lab.
Maternal immune response | Second trimester (between 22-24 weeks gestational age)
  Responses of maternal immune system advanced oxidation protein products (AOPP)) measured in chloramine units per gram of protein (micromol/g) obtained by blood withdrawal and measured in the lab.
Maternal immune response | Third trimester (between 30-32 weeks gestational age)
  Responses of maternal immune system advanced oxidation protein products (AOPP)) measured in chloramine units per gram of protein (micromol/g) obtained by blood withdrawal and measured in the lab.
Maternal immune response | Antepartum (during delivery)
  Responses of maternal immune system advanced oxidation protein products (AOPP)) measured in chloramine units per gram of protein (micromol/g) obtained by blood withdrawal and measured in the lab.
Maternal immune response | Postpartum (6-8 weeks post delivery)
  Responses of maternal immune system advanced oxidation protein products (AOPP)) measured in chloramine units per gram of protein (micromol/g) obtained by blood withdrawal and measured in the lab.
Maternal immune response | Preconceptional (up to 1 year before pregnancy)
  Tumor necrosis factor-alpha (TNF-alpha) measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | First trimester (between 7-12 weeks gestational age)
  Tumor necrosis factor-alpha (TNF-alpha) measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Second trimester (between 22-24 weeks gestational age)
  Tumor necrosis factor-alpha (TNF-alpha) measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Third trimester (between 30-32 weeks gestational age)
  Tumor necrosis factor-alpha (TNF-alpha) measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Antepartum (during delivery)
  Tumor necrosis factor-alpha (TNF-alpha) measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Postpartum (6-8 weeks post delivery)
  Tumor necrosis factor-alpha (TNF-alpha) measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Preconceptional (up to 1 year before pregnancy)
  Interleukin-6 (IL-6), measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | First trimester (between 7-12 weeks gestational age)
  Interleukin-6 (IL-6), measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Second trimester (between 22-24 weeks gestational age)
  Interleukin-6 (IL-6), measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Third trimester (between 30-32 weeks gestational age)
  Interleukin-6 (IL-6), measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Antepartum (during delivery)
  Interleukin-6 (IL-6), measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Postpartum (6-8 weeks post delivery)
  Interleukin-6 (IL-6), measured in picograms per milliliter, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Preconceptional (up to 1 year before pregnancy)
  high sensitive C-reactive protein(hsCRP), measured in mg/L, obtained by blood withdrawal and measured in the lab.
Maternal immune response | First trimester (between 7-12 weeks gestational age)
  high sensitive C-reactive protein(hsCRP), measured in mg/L, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Second trimester (between 22-24 weeks gestational age)
  high sensitive C-reactive protein(hsCRP), measured in mg/L, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Third trimester (between 30-32 weeks gestational age)
  high sensitive C-reactive protein(hsCRP), measured in mg/L, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Antepartum (during delivery)
  high sensitive C-reactive protein(hsCRP), measured in mg/L, obtained by blood withdrawal and measured in the lab.
Maternal immune response | Postpartum (6-8 weeks post delivery)
  high sensitive C-reactive protein(hsCRP), measured in mg/L, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Preconceptional (up to 1 year before pregnancy)
  Markers of the one-carbon metabolism; folate, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | First trimester (between 7-12 weeks gestational age)
  Markers of the one-carbon metabolism; folate, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Second trimester (between 22-24 weeks gestational age)
  Markers of the one-carbon metabolism; folate, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Third trimester (between 30-32 weeks gestational age)
  Markers of the one-carbon metabolism; folate, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Antepartum (during delivery)
  Markers of the one-carbon metabolism; folate, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Postpartum (6-8 weeks post delivery)
  Markers of the one-carbon metabolism; folate, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Preconceptional (up to 1 year before pregnancy)
  Markers of the one-carbon metabolism; Homocysteine, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | First trimester (between 7-12 weeks gestational age)
  Markers of the one-carbon metabolism; Homocysteine, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Second trimester (between 22-24 weeks gestational age)
  Markers of the one-carbon metabolism; Homocysteine, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Third trimester (between 30-32 weeks gestational age)
  Markers of the one-carbon metabolism; Homocysteine, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Antepartum (during delivery)
  Markers of the one-carbon metabolism; Homocysteine, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Postpartum (6-8 weeks post delivery)
  Markers of the one-carbon metabolism; Homocysteine, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Preconceptional (up to 1 year before pregnancy)
  Markers of the one-carbon metabolism; B-vitamin 12, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | First trimester (between 7-12 weeks gestational age)
  Markers of the one-carbon metabolism; B-vitamin 12, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Second trimester (between 22-24 weeks gestational age)
  Markers of the one-carbon metabolism; B-vitamin 12, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Third trimester (between 30-32 weeks gestational age)
  Markers of the one-carbon metabolism; B-vitamin 12, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Antepartum (during delivery)
  Markers of the one-carbon metabolism; B-vitamin 12, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Maternal metabolic response | Postpartum (6-8 weeks post delivery)
  Markers of the one-carbon metabolism; B-vitamin 12, measured in micromol/l, obtained by blood withdrawal and measured in the lab.
Clinical maternal outcome: gestational age | Durante partum
  Gestational age (amenorrhea duration) at delivery.
Clinical maternal outcome: pre-eclampsia | from 20 weeks of gestation to <8 weeks postpartum
  Pre-eclampsia is defined as the combination of gestational hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg (Korotkoff V) occurring after 20 weeks of gestation gestational age, measured twice, in a woman who previously had normal blood pressure) with proteinuria (≥ 300 mg/24 hours).
Clinical maternal outcome: hypertension | from 20 weeks of gestation to <8 weeks postpartum
  Hypertension is defined as a systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg (Korotkoff V) occurring after 20 weeks of gestation gestational age, measured twice, in a woman who previously had normal blood pressure.
Clinical maternal outcome: gestational diabetes | From the first positive pregnancy test to delivery
  Gestational diabetes defined as any form of hyperglycaemia detected during pregnancy, regardless ofwhether this abnormality disappears after pregnancy. Diagnosed through a 75 gr Oral Glucose Tolerance Test (OGTT) with a fasting venous value > 7 mmol/l or above 7.8 mmol/l after 2 hours.
Fetal growth | First trimester (Between 7-7+6 days of gestational age)
  Fetal growth trajectories, Crown-Rump-Length (CRL) obtained by using ultrasound imaging.
Fetal growth | First trimester (Between 9-9+6 days of gestational age)
  Fetal growth trajectories, Crown-Rump-Length (CRL) obtained by using ultrasound imaging.
Fetal growth | First trimester (Between 11-11+6 days of gestational age)
  Fetal growth trajectories, Crown-Rump-Length (CRL) obtained by using ultrasound imaging.
Fetal growth | Second trimester (Between AD 22-25 weeks of gestational age)
  Fetal growth trajectories defined as Estimated Fetal Weight (EFW) (in grams) based on the measurements (in mm) of the Head circumference (HC), Biparietal diameter (BPD), Abdominal circumference (AC) and Femur length (FL) to be obtained/measured during the ultrasound.
Fetal growth | Third trimester (Between 30-33 weeks of gestational age)
  Fetal growth trajectories defined as Estimated Fetal Weight (EFW) (in grams) based on the measurements (in mm) of the Head circumference (HC), Biparietal diameter (BPD), Abdominal circumference (AC) and Femur length (FL) to be obtained/measured during the ultrasound.
Histological placental function | Postpartum (<2 days postpartum)
  Histology of placenta: biopsies are taken within 2 days after delivery, these are snapfrozen in -80 degrees Celsius and assessed according to protocol by pathologist
Placental weight | Postpartum (<2 days postpartum)
  Placental weight measured (in grams), weighed on the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rousian M, Schoenmakers S, Eggink AJ, Gootjes DV, Koning AHJ, Koster MPH, Mulders AGMGJ, Baart EB, Reiss IKM, Laven JSE, Steegers EAP, Steegers-Theunissen RPM. Cohort Profile Update: the Rotterdam Periconceptional Cohort and embryonic and fetal measurements using 3D ultrasound and virtual reality techniques. Int J Epidemiol. 2021 Nov 10;50(5):1426-1427l. doi: 10.1093/ije/dyab030. No abstract available. PMID 34097026
- [Background] Gaillard R, Durmus B, Hofman A, Mackenbach JP, Steegers EA, Jaddoe VW. Risk factors and outcomes of maternal obesity and excessive weight gain during pregnancy. Obesity (Silver Spring). 2013 May;21(5):1046-55. doi: 10.1002/oby.20088. PMID 23784909
- [Background] Mission JF, Marshall NE, Caughey AB. Pregnancy risks associated with obesity. Obstet Gynecol Clin North Am. 2015 Jun;42(2):335-53. doi: 10.1016/j.ogc.2015.01.008. PMID 26002170
- [Background] Singh AS, Mulder C, Twisk JW, van Mechelen W, Chinapaw MJ. Tracking of childhood overweight into adulthood: a systematic review of the literature. Obes Rev. 2008 Sep;9(5):474-88. doi: 10.1111/j.1467-789X.2008.00475.x. Epub 2008 Mar 5. PMID 18331423
- [Background] Tanvig M. Offspring body size and metabolic profile - effects of lifestyle intervention in obese pregnant women. Dan Med J. 2014 Jul;61(7):B4893. PMID 25123127
- [Background] Kuhle S, Muir A, Woolcott CG, Brown MM, McDonald SD, Abdolell M, Dodds L. Maternal pre-pregnancy obesity and health care utilization and costs in the offspring. Int J Obes (Lond). 2019 Apr;43(4):735-743. doi: 10.1038/s41366-018-0149-3. Epub 2018 Jul 13. PMID 30006584
- [Background] Morgan KL, Rahman MA, Macey S, Atkinson MD, Hill RA, Khanom A, Paranjothy S, Husain MJ, Brophy ST. Obesity in pregnancy: a retrospective prevalence-based study on health service utilisation and costs on the NHS. BMJ Open. 2014 Feb 27;4(2):e003983. doi: 10.1136/bmjopen-2013-003983. PMID 24578535
- [Background] Elderman M, Hugenholtz F, Belzer C, Boekschoten M, de Haan B, de Vos P, Faas M. Changes in intestinal gene expression and microbiota composition during late pregnancy are mouse strain dependent. Sci Rep. 2018 Jul 3;8(1):10001. doi: 10.1038/s41598-018-28292-2. PMID 29968760
- [Background] Schoenmakers S, Steegers-Theunissen R, Faas M. The matter of the reproductive microbiome. Obstet Med. 2019 Sep;12(3):107-115. doi: 10.1177/1753495X18775899. Epub 2018 May 17. PMID 31523266
- [Background] Turnbaugh PJ, Hamady M, Yatsunenko T, Cantarel BL, Duncan A, Ley RE, Sogin ML, Jones WJ, Roe BA, Affourtit JP, Egholm M, Henrissat B, Heath AC, Knight R, Gordon JI. A core gut microbiome in obese and lean twins. Nature. 2009 Jan 22;457(7228):480-4. doi: 10.1038/nature07540. Epub 2008 Nov 30. PMID 19043404
- [Derived] Schenkelaars N, Wekema L, Faas MM, Steegers-Theunissen RPM, Schoenmakers S. Protocol of the PROMOTE study: characterization of the microbiome, the immune response, and one-carbon metabolism in preconceptional and pregnant women with and without obesity (an observational subcohort of the Rotterdam Periconception cohort). PLoS One. 2025 Apr 2;20(4):e0319618. doi: 10.1371/journal.pone.0319618. eCollection 2025. PMID 40173397

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT05754645/Prot_SAP_000.pdf